CLINICAL TRIAL: NCT05989360
Title: The Utility of Lung Clearance Index in Ethnic Groups and in Disease
Acronym: LUCI-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 273069
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Healthy Children; Bronchiectasis Adult; Lung Clearance Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- observational (Experimental)
  Interventions: Diagnostic Test: Lung Clearance Index

INTERVENTIONS:
Diagnostic Test: Lung Clearance Index — Normative values in healthy children from ethnic backgrounds

SUMMARY:
Introduction:

Non-CF, non-PCD bronchiectasis in children is a chronic, suppurative lung disease diagnosed by high resolution computed tomography (HRCT) imaging of the lungs. Spirometry can be abnormal in bronchiectasis but has been shown to be insensitive to early disease in other related conditions such as cystic fibrosis. Lung clearance index (LCI) could have a role in assessment of the disease.

Lung clearance index is calculated from multiple breath washout tests. There are limited data on the normative values expected using some devices, in a range of ages, and between ethnic groups.

The investigators aim to establish normative values in children aged between 6 years and 12 years, to investigate differences between ethnic groups, and to establish the relationship between lung clearance index and other measures of disease in children with bronchiectasis.

Methods:

Healthy children will be recruited from a range of settings and reviewed to ensure no previous lung disease. Children with bronchiectasis diagnosed on HRCT will be recruited from the outpatient service of Birmingham Children's Hospital.

All participants will perform lung function tests including LCI and spirometry. Basic demographic data was collected.

DETAILED DESCRIPTION:
Rationale / Hypothesis:

Hypothesis 1

Having established normative ranges helps support interpretation of lung function testing which is key to their value as an investigation. With LCI, it is important to understand the difference that may be expected between children

of different ethnic backgrounds (as demonstrated with other, non-LCI measures of lung function, where important differences between different ethnic groups has been found).

LCI is calculated from an internally adjusted measure of an individual subject's lung volume, therefore potentially negating inherent differences in ethnic variation.

Therefore we hypothesize that there are no differences in LCI in healthy children from differing ethnic backgrounds.

Evidence supporting this hypothesis is not only of intellectual value, but it would also allow clinicians to confidently interpret a range of LCI readings using globally acquired normal values. Should the data not support the hypothesis, an important direction for future research would be established.

Hypothesis 2

LCI has been demonstrated to detect small differences in lung function and correlates well with CT imaging in some disease states. There is a paucity of data in its use in its lung disease outside of CF. Current availability of easy to use, repeatable and reliable devices allows LCI to be measured in the clinic setting (Downing et al. 2016).

Understanding the relationship between CT changes and LCI in younger children with lung disease, would allow a non-invasive investigation (LCI) to be used to guide care and monitor treatment.

In order to understand how LCI changes, we also intend to determine how LCI varies in children with Non-CF, Non-PCD Bronchiectasis over a prolonged period of time.

The investigators hypothesize that in younger children with Non-CF, Non-PCD Bronchiectasis and evidence of milder disease on CT, LCI is a more sensitive disease marker than FEV1, and varies over time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children

Exclusion Criteria:

* Those with underlying respiratory/systemic disease/ prematurity

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Normative values in healthy children | 24 months
  The normative range of measurements of lung clearance index will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Nagakumar, MD, Principal Investigator — Birmingham Women's and Children's Hospital
Locations (1):
- Birmingham Children's Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No